| Mean (SD) OSDI Score | Pre | | | Post | |
|---|---|---|---|---|---|
| AS | 74.69 | | 27.72 | 27.72 | |
| PFAT+COE | 79.70 | | 37.30 | 37.30 | |
| P value | | | | | |
| Between pre-post* | p<0.0001 | | | | |
| BetweenAS- | p=0.197 p=0.199 | | | p=0.004 p=0.006 | |
| PFAT+COE** | | | | | |
| *Student's paired samples | t-test ** Independen | t samples Student's t- | test | | |
| Mean TBUT | Right eyes | Left eyes | Right | eyes | Left eyes |
| AS | 4.38 | 4.44 | 5.50 | | 5.94 |
| PFAT+ COE | 3.83 | 4.11 | 7.11 | | 6.88 |
| P value | | L | I | | 1 |
| Between pre-post* | p<0.001(right eyes) p<0.001(left eyes) | | | | |
| BetweenAS- | p=0.121 | p=0.345 | p=0.0 | p=0.04 p=0.034 | |
| PFAT+COE** | | | | | |
| *Student's paired samples | t-test ** Independen | t samples Student's t- | test | | |
| Median with | | | | | |
| interquartile range | | | | | |
| (IQR) OXFORD | | | | | |
| AS | 2(9) | | | 1(18) | |
| PFAT+COE | 2(7) | | | 1(14) | |
| P value | | | | | |
| Between pre-post* | p<0.0001 | | | | |
| BetweenAS- | p=0.366 | | | 96 | |
| PFAT+COE** | | | | | |
| *Wilcoxon signed-rank test **Mann–Whitney U test | | | | | |
| Mean Schirmer's test | Right eyes | Left eyes | Right | eyes | Left eyes |
| Result | | | | | |
| AS | 6.77 | 5.94 | 8.83 | | 9.55 |
| PFAT+COE | 6.33 | 6.33 | 18 | | 18.83 |
| P value | | 1 | | | I |
| Between pre-post* | p<0.0001(right) p<0.0001 | | | | |
| BetweenAS- | p=0.620 | p=0.593 | p<0.0 | 001 | p<0.0001 |
| PFAT+COE** | | | | | |
| *Student's paired samples t-test ** Independent samples Student's t-test | | | | | |